CLINICAL TRIAL: NCT01922154
Title: Intravitreous Ranibizumab as Adjunctive Treatment for Trabeculectomy in Neovascular Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Naris Kitnarong, Associate professor, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK002
Record Dates: First submitted 2013-08-04; First posted 2013-08-14 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Glaucoma, Neovascular
Keywords: Angiogenesis inhibitors; Neovascular; Intraocular pressure; Retinal Vein Occlusion; Vascular Endothelial Growth Factor
MeSH Terms: conditions — Glaucoma, Neovascular; Retinal Vein Occlusion | interventions — Ranibizumab; Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intravitreal ranibizumab (Experimental): Ranibizumab was injected into vitreous cavity in the study eye once (0.5 mg/0.05 ml) at least 1 week before performing trabeculectomy with mitomycin C.
  Interventions: Drug: intravitreal ranibizumab; Procedure: Trabeculectomy with mitomycinC

INTERVENTIONS:
Drug: intravitreal ranibizumab — The patients received IVR (0.5 mg in 0.05 ml) injection through the pars plana in the operating room. A fornix-based conjunctival flap technique trabeculectomy with intraoperative mitomycin C was performed within 2 weeks after IVR.
  Other Names: Lucentis; Genentech Inc, San Francisco, CA
Procedure: Trabeculectomy with mitomycinC — All participant underwent trabeculectomy with mitomycinC , which is the standard procedure for refractory glaucoma.

SUMMARY:
To evaluate the effects of intravitreal ranibizumab (IVR) as adjunctive treatment for trabeculectomy with mitomycin C (TMC) in neovascular glaucoma (NVG).

DETAILED DESCRIPTION:
This is a prospective study of 15 consecutive eyes from 14 patients (One patients had NVG in both eyes at presentation.) with NVG presented at the Department of Ophthalmology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand between December 2008 and December 2009. Each eye received IVR (0.5 mg/0.05 ml) 1 week before TMC. Trabeculectomy was performed with fornix-based conjunctival flap method.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with neovascular glaucoma
* Age more than 80 year old
* Provide written informed consent

Exclusion Criteria:

* Un-cooperated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The change of intraocular pressure (IOP) | Change of IOP between before trabeculectomy and at last visit
  The change of intraocular pressure (IOP)between before trabeculectomy with mitomycin C (TMC) and after TMC. We compared this change at several time points such as at 6, 12 months and at last visit. The most important is the change of IOP between before TMC and at last visit as well as the level of IOP at last visit which is at of the longest follow-up time.

SECONDARY OUTCOMES:
The safety of intravitreal ranibizumab (IVR) | On the day patient receives IVR
  Blood pressure (mmHg) change

CONTACTS AND LOCATIONS:
Overall Officials: Naris Kitnarong, M.D., Principal Investigator — Mahidol University
Locations (1):
- Naris Kitnarong, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitnarong N, Chindasub P, Metheetrairut A. Surgical outcome of intravitreal bevacizumab and filtration surgery in neovascular glaucoma. Adv Ther. 2008 May;25(5):438-43. doi: 10.1007/s12325-008-0047-5. PMID 18425438
- [Background] Alkawas AA, Shahien EA, Hussein AM. Management of neovascular glaucoma with panretinal photocoagulation, intravitreal bevacizumab, and subsequent trabeculectomy with mitomycin C. J Glaucoma. 2010 Dec;19(9):622-6. doi: 10.1097/IJG.0b013e3181ccb794. PMID 20179624
- [Result] Dunavoelgyi R, Zehetmayer M, Simader C, Schmidt-Erfurth U. Rapid improvement of radiation-induced neovascular glaucoma and exudative retinal detachment after a single intravitreal ranibizumab injection. Clin Exp Ophthalmol. 2007 Dec;35(9):878-80. doi: 10.1111/j.1442-9071.2007.01632.x. PMID 18173426